CLINICAL TRIAL: NCT01455701
Title: A Phase I Pharmacokinetic and Safety Study of Tocilizumab (TCZ) in Patients Less Than 2 Years Old With Active Systemic Juvenile Idiopathic Arthritis (sJIA)
Brief Title: A Study to Evaluate Pharmacokinetics and Safety of Tocilizumab (RoActemra/Actemra) in Participants Less Than 2 Years Old With Active Systemic Juvenile Idiopathic Arthritis (sJIA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25737; 2015-000435-33 (EudraCT Number)
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab intravenous (IV) infusion at a dose of 12 milligrams per kilogram (mg/kg) every two weeks (Q2W) during main evaluation period of 12 weeks (a total of 6 infusions including one at baseline visit). Participants will have the option to be treated in an optional extension period after completion of main evaluation period. In optional extension period, participants will receive tocilizumab 12 mg/kg IV infusion Q2W from Week 12 until the participant reaches 2 years of age or has been treated for one year from baseline, whichever is longer.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered as indicated in the arm description.
  Other Names: RoActemra; Actemra; RO4877533

SUMMARY:
This is a multi-center, open-label single-arm study to investigate the pharmacokinetics and safety of tocilizumab (RoActemra/Actemra) in participants less than 2 years old with active sJIA. Participants will receive tocilizumab infusions every 2 weeks. The anticipated time on study treatment is 12 weeks (Main evaluation period). Participants will have the option to continue tocilizumab treatment until participant reaches 2 years of age or up to one year from baseline, whichever is longer. An optional extension period will follow the main evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Fulfils international league of associations for rheumatology (ILAR) classification criteria for sJIA
* Duration of sJIA symptoms lasting for at least 1 months subsequent to diagnosis of sJIA
* Presence of active disease as determined by the presence of:

  1. Greater than or equal to (>=) 2 active joints at screening and baseline, with at least 14 consecutive days of temperature recordings, which may include the presence or absence of fever (>=38 degree Celsius) during the time between screening and baseline; or
  2. >=2 active joints at screening and baseline, with a fever >=38 degree Celsius for at least 5 consecutive days during the time between screening and baseline; under these circumstances a participant does not need to complete a full 14 days of temperature diary entries to meet this inclusion criteria
* Not currently receiving corticosteroids (CS) or if taking oral CS like prednisone or equivalent, the dose should be less than or equal to (<=) 1 milligram per kilogram per day (mg/kg/day) and the dose has remained stable for at least 2 weeks prior to baseline
* Not currently receiving methotrexate (MTX) or if taking MTX (together with either folic acid or folinic acid according to local standard-of-care), the dose has remained stable or has been discontinued for at least 4 weeks prior to baseline
* Not currently receiving non-steroidal anti-inflammatory drugs (NSAIDs) or if taking NSAID, the dose has remained stable or has been discontinued for at least 2 weeks prior to baseline
* If the participants has received previous treatment with any of the following biologic agents, these must have been discontinued according to the following timelines prior to the baseline visit and are not permitted during the study:

  1. Etanercept must have been discontinued within >= 2 weeks prior to baseline
  2. Anakinra must have been discontinued within >= 4 days prior to baseline
  3. Abatacept must have been discontinued within >= 12 weeks prior to baseline
  4. Infliximab or adalimumab must have been discontinued within >= 8 weeks prior to baseline
  5. Canakinumab must have been discontinued within >= 20 weeks prior to baseline
  6. Rilonacept must have been discontinued within >= 6 weeks prior to baseline
  7. Golimumab must have been discontinued within >= 10 weeks prior to baseline
  8. Certrolizumab pegol must have been discontinued within >= 10 weeks prior to baseline
* History of inadequate clinical response (in the opinion of the treating physician) to NSAIDs and CS

Exclusion Criteria:

General Exclusion Criteria:

* Any autoimmune, rheumatic disease or overlap syndrome other than sJIA
* Not fully recovered from recent surgery or less than 6 weeks since surgery, at the time of screening visit; or planned surgery during the study (except for myringotomy surgery, which is permitted)

General Safety Exclusion Criteria:

* Any significant concurrent medical or surgical condition which would jeopardize the participant's safety or ability to complete the trial
* History of significant allergic or infusion reactions to prior biologic therapy or to any of the excipients listed in tocilizumab product labelling documents
* Inborn conditions characterized by a compromised immune system
* Known human immunodeficiency virus (HIV) infection or other acquired forms of immune compromise
* Evidence of serious uncontrolled concomitant diseases including but not limited to the nervous system, renal, hepatic or endocrine systems
* Asthma for which the participant has required the use of oral or parenteral corticosteroids for >=2 weeks within 6 months prior to baseline visit
* Any active acute, subacute, chronic or recurrent bacterial, viral or systemic fungal infection
* History of atypical tuberculosis (TB)
* Active TB requiring treatment at any point prior to screening visit
* Positive TB test result at screen, unless treated with anti-TB therapy for at least 4 weeks prior to receiving study medication and chest radiograph is negative for active TB within 6 months of screening visit consistent with local practice
* Any major episode of infection requiring hospitalization or treatment during screening or treatment with IV antibiotics completing within 4 weeks of the screening visit or oral antibiotics completing within 2 weeks of the screening visit
* History of reactivation or new onset of a systemic infection such as herpes zoster or Epstein Barr virus within 2 months of the screening visit
* History of hepatitis B or hepatitis C infection
* Chronic hepatitis - viral or autoimmune
* Significant cardiac or pulmonary disease
* History or concurrent serious gastrointestinal disorders such as ulcer or inflammatory bowel disease, ulcerative colitis or other symptomatic lower gastrointestinal conditions, including ulcer and perforation
* History of or current cancer or lymphoma
* History of macrophage activation syndrome (MAS) within 3 months prior to the screening visit
* Uncontrolled diabetes mellitus with elevated hemoglobin A1c (HbA1c) as defined by age-specific standards

Excluded Previous or Concomitant Therapy:

* Participation in another interventional clinical trial within the past 30 days or 5 serum half-lives of the investigative medication, whichever is longer
* Previous treatment with tocilizumab
* Administration of IV immunoglobulin within 4 weeks prior to the baseline visit
* Previous treatment with any cell depleting therapies, including investigational agents
* Prior stem cell transplant at any time
* Live or attenuated vaccines within 4 weeks prior to the baseline visit, or intending to receive while on study medication or 8 weeks following the last dose of study medication
* Serum creatinine >1.5 ULN (upper limit of normal for age and sex)
* AST or ALT > 1.5 ULN (upper limit of normal for age and sex)
* Total bilirubin > 1.3 mg/dL (> 23 umol/L)
* Platelet count < 200 x103/μL (< 200,000/mm3)
* Hemoglobin < 7.0 g/dL (< 4.3 mmol/L)
* WBC count < 6,200/mm3 (< 6.2 x 109/L)
* Neutrophil count < 2,500/ mm3 (< 2.5x 109/L)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Tocilizumab | Pre-infusion (Hour 0) on Days 1, 15, 29, 43, 57, 71, and 85; at the end of infusion on Days 1, 29 and 71; and anytime on Days 8, 36, and 78 (infusion length = 1 hour)
  Pharmacokinetic profile of tocilizumab is evaluated in terms of model predicted Cmax at steady state. Pharmacokinetic-evaluable population includes all participants who provided at least one serum pharmacokinetic sample with valid concentration data.
Minimum Serum Concentration (Cmin) of Tocilizumab | Pre-infusion (Hour 0) on Days 1, 15, 29, 43, 57, 71, and 85; at the end of infusion on Days 1, 29 and 71; and anytime on Days 8, 36, and 78 (infusion length = 1 hour)
  Pharmacokinetic profile of tocilizumab is evaluated in terms of observed Cmin at day 85. Pharmacokinetic-evaluable population.
Model predicted Area Under the Serum Concentration-Time Curve from Time Zero to End of Dosing (AUCtau) of Tocilizumab | Pre-infusion (Hour 0) on Days 1, 15, 29, 43, 57, 71, and 85; at the end of infusion on Days 1, 29 and 71; and anytime on Days 8, 36, and 78 (infusion length = 1 hour)
  AUCtau is the model-predicted area under the tocilizumab serum concentration versus time curve from time zero to the end of dosing interval (2 weeks). Pharmacokinetic-evaluable population.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs | Baseline up to end of the study (up to approximately 60 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (9):
  - Children's National Medical Center; Pediatric Rheumatology, Washington D.C., District of Columbia
  - The University of Chicago;Department of Pediatrics, Chicago, Illinois
  - University of Louisville Research Foundation, Inc; Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - The Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Children's Hospital Boston Pediatric Medicine, Boston, Massachusetts
  - Children's Speciality Center of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center; Pediatric Rheumatology, Hackensack, New Jersey
  - Cincinnati Children'S Hospital Medical Center; Division of Rheumatology, Cincinnati, Ohio
  - Children's Hospital Of Pittsburgh, Pittsburgh, Pennsylvania
- Hospital Gral de Niños Pedro Elizalde, Buenos Aires, Argentina
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (3):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Hospital For Sick Children, Toronto, Ontario
  - McGill University; Montreal Children's Hospital; Inflammatory, Autoimmune & Bone, Montreal, Quebec
- Klinik Bremen-Mitte; Prof. Hess-Kinderklinik, Bremen, Germany
- Semmelweis University; 2nd Department of Paediatrics, Budapest, Hungary
- Poland (2):
  - Uniwersytecki Szpital Kliniczny Nr 4 im. M. Konopnickiej; Oddz. Kardiolog. i Reumatolog. dla Dzieci, Lodz
  - Uniwersytecki Szpital Dzieciecy w Lublinie; Oddzial Pediatrii, Chorob Pluc i Reumatologii, Lublin
- Hospital Universitario la Fe: Servicio de Reumatologia Pediatrica, Valencia, Spain

REFERENCES:
- [Derived] Mallalieu NL, Wimalasundera S, Hsu JC, Douglass W, Wells C, Penades IC, Cuttica R, Huppertz HI, Joos R, Kimura Y, Milojevic D, Rosenkranz M, Schikler K, Constantin T, Wouters C. Intravenous dosing of tocilizumab in patients younger than two years of age with systemic juvenile idiopathic arthritis: results from an open-label phase 1 clinical trial. Pediatr Rheumatol Online J. 2019 Aug 22;17(1):57. doi: 10.1186/s12969-019-0364-z. PMID 31438986